CLINICAL TRIAL: NCT07042243
Title: The Florida Partnership for Adding Social Context to Address Cancer Survivorship Outcomes (Florida ASCENT)
Brief Title: The Florida ASCENT Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB202500820; PRO00064441 (Other Grant/Funding Number: FL DEPT OF HLTH)
Record Dates: First submitted 2025-06-09; First posted 2025-06-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Food Deprivation; Food Habits; Food Selection; Colorectal Cancer; Prostate Cancer; Lung Cancer; Breast Cancer; Gynecologic Cancer; Hematologic Cancer; Skin Cancer; Melanoma; Nutrition Poor; Nutritional Deficiency
Keywords: Food Insecurity; Cancer; Food Access; Community-Informed Research; Nutritional Needs; Mixed-Methods
MeSH Terms: conditions — Neoplasms; Feeding Behavior; Food Preferences; Colorectal Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Breast Neoplasms; Hematologic Neoplasms; Skin Neoplasms; Melanoma; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Access to the randomization list will be given only to project staff not involved in participant screening and enrollment to ensure objectivity and blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving Standard care and MyCarePulse (No Intervention): Participants not receiving the ASCENT Patient Navigator intervention, but are still utilizing MyCarePulse for comparison purposes. This arm will be conducted in phase 2 of the study and will have 50 participants (25 per site).
- Participants receiving ASCENT Patient Navigator (PN) Intervention and MyCarePulse (Experimental): Participants will be receiving the ASCENT Patient Navigator intervention, and the MyCarePulse tool will flag participants who need assistance. They will then be connected to an ASCENT Patient Navigator to get those needs assessed. This arm will be conducted in phase 2 of the study and will have 50 participants (25 per site).
  Interventions: Behavioral: MyCarePulse and ASCENT PN

INTERVENTIONS:
Behavioral: MyCarePulse and ASCENT PN — The combination of a digital platform and patient navigators assisting the process. Also, taking a multi-level approach engaging community members, patients, and providers in phase one through qualitative interviews. Then using the findings to adapt MyCarePulse for the clincial trial in phase two.
  Arms: Participants receiving ASCENT Patient Navigator (PN) Intervention and MyCarePulse

SUMMARY:
The goal of this clinical trial is to adapt, implement, and evaluate MyCarePulse and ASCENT patient navigator to overcome barriers to care among patients with cancer.

The main hypotheses it aims to test are:

* At the patient level, the intervention will result in higher levels of food security, self- efficacy for dietary behaviors, and higher diet quality than standard care.
* At the provider level, the intervention will be feasible, acceptable, appropriate, and able to enhance individualized care for patient wellness.

Researchers will compare cancer patients receiving the MyCarePulse and ASCENT patient navigator intervention to those receiving standard care, to see if the intervention improves food security, self-efficacy, and diet quality.

Phase 1

Patient Participants will:

* Complete the ASCENT Questionnaire, which is comprised of the following:

  * U.S. Food Security Survey Module (U.S. FSSM)
  * Patient-Reported Outcomes Measurement Information System (PROMIS-29)
  * Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
* Be assessed using the Veggie Meter instrument
* Participate in two semi-structured interviews

Provider Participants will:

•Participate in one semi-structured interview

Phase 2

Patient Participants will:

* Participate in ASCENT patient navigator screenings and consultations
* Complete the ASCENT Questionnaire, which comprises the U.S. FSSM, PROMIS-29, and ASA24®

DETAILED DESCRIPTION:
This study aims to establish a clinical trial of 200 cancer patients at the UF Health and University of Miami Health Systems (100 in Phase 1 and 100 in Phase 2). UF Health will serve as the Coordinating Center for the study.

Building on My Wellness Check, an electronic health records (EHR)-based referral system developed at the University of Miami for symptom and practical needs screening in cancer patients. This study will integrate the platform with a network of patient navigators who can provide individualized support and connect survivors with relevant community resources to promote healthy eating under a program called MyCarePulse.

The main objective is to adapt, implement, and evaluate MyCarePulse and ASCENT patient navigator to overcome barriers to care among patients with colorectal, prostate, lung, breast, gynecologic, hematologic, and skin (including melanoma) cancers

This study will take place in two phases. Phase 1 will consist of implementation strategy and Phase 2 will consist of the intervention phase.

Phase 1 has two aims:

In Aim 1, we will test the hypothesis that the ASCENT intervention, delivered through the MyCarePulse Research Portal, is implemented as intended using community-engaged participatory design methods to refine multilevel approaches.

In Aim 2, we will build readiness for the implementation of the MyCarePulse Research Portal and ASCENT patient navigator using the Expert Recommendations for Implementing Change (ERIC) strategies.

Phase 2 has one aim:

In Aim 3, we will implement and evaluate MyCarePulse Research Portal and ASCENT patient navigator in a randomized trial.

ELIGIBILITY:
Patient Eligibility Inclusion Criteria:

1. ≥18 years old.
2. Pathologically confirmed diagnosis of colorectal, prostate, lung, breast, gynecologic, hematologic, or skin (including melanoma) cancer within the past 12 months.
3. Self-reported ability to read and speak English.
4. Able to provide informed consent.
5. Participant must not be considered a "vulnerable population" (pregnant women, neonates, children etc.)

Patient Eligibility Exclusion Criteria:

1. ≤18 years old.
2. Participant do not have a pathologically confirmed diagnosis of colorectal, prostate, lung, breast, gynecologic, hematologic, or skin (including melanoma) cancer within the past 12 months.
3. Participant does not live within the state of Florida.

3) Does not self-reported ability to read and speak English or Spanish. 4) Not able to provide informed consent. 5) Participant is considered a "vulnerable population" (pregnant women, neonates, children etc.)

Provider Eligibility Inclusion Criteria

1. ≥18 years old.
2. Currently works as a physician, physician assistant, patient navigator and/or health system/administrative leader in UF and UM affiliated clinics.
3. Self-reported ability to read and speak English or Spanish.
4. Able to provide informed consent.
5. Participant must not be considered a "vulnerable population" (pregnant women, neonates, children etc.)

Provider Eligibility Exclusion Criteria

1. ≤ 18 years old.
2. Does not currently works as a physician, physician assistant, patient navigator and/or health system/administrative leader in UF and UM affiliated clinics.
3. Does not self-report having the ability to read and speak English.
4. Not able to provide informed consent.
5. Participant is considered a "vulnerable population" (pregnant women, neonates, children etc.)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Food security from Baseline using U.S. FSSM | 6 months
  Self-reported by patient using the US Food Security Module (US FSSM). The US FSSM consists of 18 questions for homes with children under the age of 18 years and 10 items for households without children, e.g., a query regarding the use of emergency foods from food banks, soup kitchens, or other organizations by household members within the past year. The overall food security status (full, marginal, low and very low) will be determined by the number of affirmative responses to those questions.
Change in Diet quality from Baseline using the ASA24 Dietary Recall Assessment and the Veggie Meter Instrument | 6 months
  Evaluated by the ASA24 dietary recall assessment and Veggie Meter Instrument. The ASA24 dietary recall collect information on calorie intake and nutrient density, and will be assessed using the Healthy Eating Index (HEI), 2015 version. The Veggie Meter Instrument will give a score from 0-800, and higher scores are associated with greater fruit and vegetable intake.
Change in Self efficacy for dietary behaviors from Baseline using the the Preferences and Self-Efficacy of Diet and Physical Activity Behaviors Scale | 6 months
  Self-reported by patient using the the Preferences and Self-Efficacy of Diet and Physical Activity Behaviors scale. The scale measures preferences and self-efficacy for four behaviors: fruit and vegetable intake, dietary fat intake, added sugar intake and physical activity. A sample question is "Did MyCarePulse make you confident to eat healthy snacks like a fruit or a vegetable when you are really hungry?"

SECONDARY OUTCOMES:
SDOH Barriers Resolution in Patient Participants using the AHC HRSN Screening Tool | Baseline and 6 months Post-Intervention
  The resolution of SDOH Barriers will be calculated from pre/post patient-reported assessments using AHC HRSN Screening Tool. The 13-item Centers for Medicare, Medicaid Services Accountable Health Communities Health-Related Social Needs (AHC HRSN) Screening Tool64. The AHC HRSN Screening Tool covers multiple dimensions of patient wellness, including diet quality, physical fitness, social support, and mental health.
Change in Health-related quality of life from Baseline using the PROMIS-29 Profile | Baseline and 6 months post-Intervention
  Determined by pre/post-intervention assessment using the Patient-Reported Outcomes Measurement Information System, PROMIS-29 Profile, to assess health-related quality of life98. The PROMIS-29 comprises 29 items that include anxiety, depression, fatigue, pain interference, sleep disturbance, physical function, and ability to participate in social roles and activities.
Change in Feasibility, acceptability, and appropriateness of the intervention using REST to measure the implementation outcomes of FIM, AIM, and IAM | Baseline and 6 months Post-Intervention
  The implementation outcomes of FIM, AIM, and IAM will be measured using the Research Engagement Survey Tool (REST). Clinical staff will complete these measures prior to patient enrollment and at the end of the study. All individuals engaged in planning or delivery of the intervention will complete it to determine the level of community engagement. Descriptive analyses will be used to characterize responses.

OTHER OUTCOMES:
Change in Organizational Readiness from Baseline using the MORE Questionnaire | Baseline and 6 months Post-Intervention
  The Measures of Organizational Readiness for Patient Engagement (MORE)83 will reflect the implementation context. It will be delivered pre- and post-intervention to assess change in organizational readiness during the ERIC adaptations and post-implementation. Clinical staff and clinic leadership to will be recruited to complete measures at the completion of in-clinic data collection periods.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States